CLINICAL TRIAL: NCT02484495
Title: Evaluate the Impact of Package of Interventions on Growth and Micronutrient Status of Infant and Young Children
Brief Title: Extended Pilot Project Community Based Production of Complementary Food in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: Micronutrient Initiative (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPHI_FSNRD_CF_MNP002
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-02

CONDITIONS: Growth Acceleration; Infant Morbidity
Keywords: Complementary feeding recommendation; Program evaluation; Process and impact evaluation
MeSH Terms: interventions — Program Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Program evaluation in intervention areas (Experimental): A quasi-experimental matched-control cluster design will be used in which outcomes are compared in intervention and non-intervention areas. The program evaluation will have three points of data collection to assess effect of the program on the nutritional status of children 6-29 months. Sixty intervention clusters have been purposively selected whereas the data will be collected from randomly selected subjects. The following interventions will be provided:
  * Processed complementary food rations will be distributed to all children 6-23 months of age, from a grain bank based on bartering of raw materials.
  * Monthly 15 sachets of MNP will be provided to all children 6-23 months of age with the instruction to add them to their complementary food, to enable point-of-use fortification.
  Interventions: Other: Program evaluation (impact assessment)
- Non intervention areas (No Intervention): A quasi-experimental matched-control cluster design will be used in which outcomes will be compared in intervention and non-intervention clusters. The program evaluation will have three points of data collection to assess effect of the program on the nutritional status of children 6-29 months. Matching sixty non-intervention clusters have been purposively selected out of the predetermined non- intervention districts whereas study subjects will be randomly selected from the identified clusters on a population based sampling method both groups. These non-intervention areas do not get processed complementary food rations and do not receive MNPs.

INTERVENTIONS:
Other: Program evaluation (impact assessment) — The program activities include: processed complementary food rations which will be distributed to all children 6-23 months of age, in a grain bank based on bartering of raw materials; enhanced Infant and Young Child Nutrition (IYCN) counselling will be given to the mothers of children 6-23 month of age, using improved Behavior messages based Change Intervention (BCI) on formative research.
  Monthly 15 MNPs sachets will be provided to all children 6-23 months of age with the instruction to add them to their complementary food, to enable point-of-use fortification on every alternate day.
  Arms: Program evaluation in intervention areas

SUMMARY:
The purpose of the study is to evaluate the impact of a package of interventions including production and distribution of locally produced complementary foods (via so-called "Grain-banks") and Micronutrient Powders (MNPs) supplementation, and optimized food based Complementary Feeding Recommendation, on growth and micronutrient status of infants and young children. The impact of the intervention package will be evaluated in a quasi-experimental matched-control cluster design in infants and young children between 6 - 29 months of age. The impact, outcome, and output indicators of infants/children will be assessed in cross-sectional samples at baseline, after 9 and 18 months. A total of60 pair clusters are selected in which 15 households per cluster will be identified from the eligible population. A total of 1800 children from intervention and match-controlled clusters, will be sampled in the target age groups. Qualitative and quantitative data will be collected to gather information on Knowledge, Attitude and Practice (KAP), Infant and Young Child Feeding practices, anthropometry and anemia, following the impact pathway developed for the study.

Research questions to be answered in this program evaluation are:

1. What impact does the extended pilot (implementation of local complementary food production and MNP) have on:

   1. Growth in children 17-29 months of age
   2. Infant and Young Child Feeding practices in children (6-23m), and
   3. Anemia status in children 11-23 m?
2. What are determining factors for the impact/no impact related to:

   1. Immediate outcomes: skills and capacity; knowledge, attitude and practices; and improved access
   2. Intermediate outcomes: utilization; provision, and ensuring enabling environment
   3. Program performance as measured by program monitoring data on output and activities?

DETAILED DESCRIPTION:
The aim of this study is to assess the impact/effectiveness of the improved interventions on infant growth and micronutrient status so as to measure what would have happened in the absence of interventions. The study will be conducted in the same four regions in Ethiopia where the program intervention is taking place namely, Amhara, Tigray, Oromiya, and South Nations Nationalities and Peoples Region (SNNPR) regions.

* Sample size calculations assume an expected difference of 0.2 Standard Deviation (SD) in HAZ, and 5% difference in feeding practices, 80% power, and α-error of 5%; and a cluster effect of approximately 2.
* A total of 1800 children will be sampled in both intervention and non-intervention (control) villages. A total of 120 clusters are chosen for both groups. Each intervention cluster will be matched with a control cluster selected to be similar in geographical and ecological conditions, access to a health-care centre, status of food security and the existence of Community Based Nutrition (CBN) programme. Within each pair of clusters, households will be randomly selected after the complete listing of eligible households. A total of 15 households will be identified in each 120 clusters.
* Demographics and socio-economic status indicators will be collected using Demographic Health Surveys (DHS) methods.
* Infant and Young Child feeding indicators will be assessed in all children 6-23 months at baseline, mid- and endline
* Knowledge attitude and practices concerning the intervention exposure indicators including perceptions and utilization of complementary food, MNP, and the use and perceptions on the grain banks will be assessed at baseline, mid- and endline in caregivers.

Data analysis include:

* For demographic and socio- economic characteristics of the study participants descriptive statistics will be used.
* To calculate the nutritional status of children 6-23 months, Epi-Info/Emergency Nutrition Action (ENA) for SMART software will be used.
* The median (min, max) of the weight or number of MNP consumed per day during the intervention period will be calculated as measure of compliance; however analyses will be done based on intention-to-treat.
* Qualitative data will be recorded in digital recorders which will be transcribed first to local language then to English. Then specific themes will be identified and matrices will be prepared and data will be analysed.
* The qualitative data will be analysed separately and triangulation will be made to compare the results.
* All analysis will be done on an intention-to-treat basis, taking into account the matched-controlled design. For continuous variables we will use linear mixed models that include cluster, household and child as random effects to account for clustered observations. Fixed effects to be included in the model are covariates such as child's sex, age, household socio-economic status and relevant baseline values. Normality will be examined by creating a Quantile-Quantile (QQ) plot and subsequent visual inspection. Equal variances will be assured with Levene's test.
* For categorical variables mixed-effects logistic regression models will be used with random effects for cluster and households.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6-23 m of age who receive Complementary Food (CF) through grain bank or commercial central production
* Living in one of the selected clusters(for intervention and nonintervention clusters)
* Those who receive MNP (15 sachets/month/child)
* Receive enhanced IYCF counselling
* Receive food based Complementary Food Recommendation (CFR)
* Free of chronic conditions that may impact their health

Exclusion criteria:

* Children between 6-23 m of age who do not get CF either through grain bank program or central production
* Those who do not get MNP
* Those who do not receive food based CFR
* Children with a chronic disease and/or chronic use of medications

Ages: 6 Months to 29 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
% of children 17-29 months of age with HAZ < -2 SD | Up to 18 months
  The ultimate outcomes of the program are improved nutritional status of children which include improved Z-scores for height-for-age (HAZ) according to the child growth standard.

SECONDARY OUTCOMES:
Mean height | Up to 18 months
  Mean Height : Measured using standardized instruments
Z score: | Up to 18 months
  Change in weight-for-length Z-score (WHZ), and weight-for-age Z-score (WAZ)
  % of wasted and underweight children Number of stunted, wasted, underweight children/Number of normal childrenX100
Morbidity | Up to 18 months
  - including incidence of acute diarrhea episodes (>3 loose stools/day)-incidence of respiratory infection episodes (cough and/or difficult breathing with or without fever, accompanied by rapid breathing and chest in drawing) in the last 2 weeks prior to the survey
Anemia status | Up to 18 months
  Hemoglobin level as measured by Hemocue and adjusted for altitude
% of children 6-23 months of age who were fed an minimum acceptable diet | Up to 18 months
  Measured using 24 hr recall method
Mean weight | Up to 18 months
  Mean weight: Measured using standardized instruments

CONTACTS AND LOCATIONS:
Overall Officials: Saskia JM Osendarp, PhD, Study Chair — Micronutrient Initiative; Inge D Brouwer, PhD, Study Director — Wageningen University
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Menon P, Rawat R, Ruel M. Bringing rigor to evaluations of large-scale programs to improve infant and young child feeding and nutrition: the evaluation designs for the Alive & Thrive initiative. Food Nutr Bull. 2013 Sep;34(3 Suppl):S195-211. doi: 10.1177/15648265130343S206. PMID 24261077
- [Background] Ton G. The Mixing of Methods: A Three-Step Process for Improving Rigour in Impact Evaluations, LEI, In: RESEARCH WUA, CENTER eds. THE NETHERLANDS.; 2012
- [Background] Kusters CSLea. Making evaluations Matter: A practical guide for evaluators. Center for Development Innovations. . In: Wageningen University and Research centre ed. Wageningen, The Netherlands; 2011
- [Background] WHO. Indicators for assessing infant and young child feeding practices. Part I definitions. 2008